CLINICAL TRIAL: NCT00322608
Title: Phase I Study of the Vascular Disrupting Agent NPI-2358 Administered Via Intravenous Infusion in Patients With Advanced Solid Tumor Malignancies or Lymphoma
Brief Title: Study of the Vascular Disrupting Agent NPI-2358 in Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nereus Pharmaceuticals, Inc. (Industry)
Responsible Party: Kristine C. Federico RN,BSN, Nereus Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI-2358-100
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Cancer
Keywords: Solid Tumors; Lymphomas
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — NPI 2358

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental)
  Interventions: Drug: NPI-2358

INTERVENTIONS:
Drug: NPI-2358 — Treatment on Days 1, 8 and 15 in a 28 day cycle

SUMMARY:
This is a Phase 1 clinical trial examining the safety, pharmacokinetics and pharmacodynamics of escalating doses of the vascular disrupting agent NPI-2358 in patients with refractory solid tumors or lymphoma. The formation of new blood vessels (angiogenesis) is an important component of tumor growth and vascular disrupting agents are intended to target the differences between these tumor blood vessels and the blood vessels in normal tissues. NPI-2358 has also been seen to directly affect tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status ≤ 2
* Pathologically or histologically confirmed solid tumor malignancy
* Patients must not be candidates for regimens known to provide clinical benefit.
* All adverse events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v. 3.0) Grade ≤ 2, except for neurological toxicity that must have resolved to Grade ≤ 1.
* Adequate bone marrow reserve, hepatic and renal function
* Signed informed consent

Exclusion Criteria:

* Administration of chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic) within 21 days prior to receipt of study medication (6 weeks for nitrosoureas or mitomycin C; 12 weeks for radioimmunotherapy). Major surgery, other than diagnostic surgery, within 6 weeks before first study drug administration. Radiotherapy within 4 weeks (some types of radiation therapy are excluded regardless of interval since treatment).
* Significant cardiac history or findings
* Underlying conditions or medications associated with bleeding diathesis
* Disorders associated with significant vascular pathology
* Lung cancer with central chest tumors
* Prior treatment with vascular disruptive agents
* Seizure disorder requiring anticonvulsant therapy; prior transient ischemic attack or cerebrovascular accident
* Brain metastases
* Severe chronic obstructive pulmonary disease (COPD) with hypoxemia
* Active uncontrolled bacterial, viral, or fungal infection, requiring systemic therapy
* Known infection with human immunodeficiency virus (HIV), active hepatitis A, B, or C
* Patients with a prior hypersensitivity reaction to any product containing Solutol and/or propylene glycol
* Pregnant or breast-feeding women. Female patients must be postmenopausal, surgically sterile or they must agree to use acceptable methods of birth control. Female patients with childbearing potential must have a negative serum pregnancy test. Male patients must be surgically sterile or agree to use an acceptable method of contraception.
* Concurrent, active second malignancy for which the patient is receiving therapy, excluding basal cell carcinoma of the skin or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety | continuously
Tolerability | continuously
Maximum tolerated dose (MTD) | continuously

SECONDARY OUTCOMES:
Pharmacokinetics | continuously
Pharmacodynamics | continuously
Response Evaluation Criteria in Solid Tumors (RECIST) | continuously

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Spear, M.D., Study Director — Chief Medical Officer, Nereus Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute/Wayne State University, Detroit, Michigan
  - Institute for Drug Development, San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington